CLINICAL TRIAL: NCT05848375
Title: Rotator Cuff Repair Under Isolated Loco-regional Anesthesia Versus General Anesthesia Combined With Loco-regional Anesthesia: Randomized Controlled Trial of Superiority.
Brief Title: Rotator Cuff Repair Under Isolated Loco-regional Anesthesia
Acronym: AGORA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-A00499-36
Record Dates: First submitted 2023-04-21; First posted 2023-05-08 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Cuff Surgical Repair
MeSH Terms: interventions — Ropivacaine; Levobupivacaine

STUDY DESIGN:
Intervention Model Description: Interventional study, randomized in two parallel groups, multicenter (trial of superiority) :
  The research procedure for arthroscopic rotator cuff repair is performed under local regional anesthesia alone without general anesthesia. LRA is performed by injecting anesthetic into the interscalene nerve block under ultrasound guidance. This LRA can be accompanied by hypnotic or morphine sedation. The comparison procedure is arthroscopic rotator cuff repair performed under LRA and GA
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loco regional anesthesia alone (Experimental): Arthroscopic rotator cuff repair performed under LRA alone
  Interventions: Procedure: Arthroscopic rotator cuff repair; Drug: naropeine or chirocaine (Arthroscopic rotator cuff repair under LRA)
- Loco regional anesthesia associated to general anesthesia (Active Comparator): Arthroscopic rotator cuff repair performed under LRA and GA
  Interventions: Procedure: Arthroscopic rotator cuff repair; Drug: naropeine or chirocaine (Arthroscopic rotator cuff repair under LRA associated to GA)

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair — The operation involves systematic acromioplasty during the supra +/- infraspinatus repair and sometimes requires a tenotomy of the long biceps if it is pathological.
Drug: naropeine or chirocaine (Arthroscopic rotator cuff repair under LRA associated to GA) — Loco Regional Anesthesia is performed by injecting anesthetic (between 10 and 20 ml of naropeine or chirocaine) into the interscalene nerve block under ultrasound guidance associated to General Anesthesia performed by injection of diprivan and ultiva.
  Arms: Loco regional anesthesia associated to general anesthesia
Drug: naropeine or chirocaine (Arthroscopic rotator cuff repair under LRA) — Loco Regional Anesthesia is performed by injecting anesthetic (between 10 and 20 ml of naropeine or chirocaine) into the interscalene nerve block under ultrasound guidance
  Arms: Loco regional anesthesia alone

SUMMARY:
Damage to the tendons of the shoulder, called rotator cuff, causes pain and loss of strength that may require surgery. This operation is performed under general anesthesia combined with loco-regional anesthesia of the shoulder. Indeed, this loco-regional anesthesia makes it possible to specifically suppress the sensation of pain in the shoulder for several hours after surgery. General anesthesia is produced by injecting drugs intravenously and breathing anesthetic vapors. Repair of the rotator cuff under loco-regional anesthesia alone is performed by several surgeons in France and is recommended by international experts. If blood pressure is artificially lowered during general anesthesia, loco-regional anesthesia alone allows maintenance of blood pressure and real-time clinical assessment since the patient is conscious.

The purpose of the research is to compare the blood pressure measured during surgery of patients operated under loco-regional anesthesia alone or associated with general anesthesia, two common practices of surgical teams.

DETAILED DESCRIPTION:
Rotator cuff injury is a common pathology with a prevalence of 30% in the general population. The main symptom of a rotator cuff tear is pain. It can be sharp when it is accidental or manifests itself when the shoulder is solicited, frequently waking the patient at night. Conservative treatment may be offered in some patients, but in the event of prolonged pain or significant lesions, surgery is recommended.

The gold standard treatment for rotator cuff tears is arthroscopic surgery. The anesthesia performed is a general anesthesia (GA) associated with a loco-regional anesthesia (LRA) of the shoulder. The injection of anesthetics into the brachial plexus before general anesthesia allows better control of postoperative pain. GA is given to patients after LRA, using a combination of hypnotic agents, curare and morphine, both for induction and maintenance of anaesthesia.

GA has several advantages: patients with a rotator cuff tear do not experience pain during surgery. For the surgeon, the GA is comfortable since the patient remains motionless throughout the duration of the surgery. Nevertheless, this requires the availability of these drugs but also increases the risk of viral contamination, mainly due to COVID-19. During the first wave of the pandemic in March 2020, several countries in Europe were in need of curare and hypnotic agents. These specific drugs for anesthesia were administered in priority to patients requiring emergency GA or for carcinological surgery. Rotator cuff tears have therefore become irreparable, due to tendon retraction or fatty infiltration into the muscle, in patients with surgery postponed for several months.

The recent development of ultrasound facilitates the realization of the LRA, allowing a better identification of the brachial plexus, for the injection of the anesthetic, resulting in a complete anesthesia of the shoulder. Even if the efficacy of LRA alone has already been described by several groups in non-GA shoulder surgeries, before 2020 it was rarely performed to repair rotator cuff tears under arthroscopy.

Rotator cuff repair under LRA alone has been performed by several surgeons in France since COVID-19 and is now recommended by international experts. Particular attention should be paid to positioning the patient, maintaining cerebral perfusion and oxygenation. Methods of measuring cerebral perfusion or oxygenation are too slow for real-time assessment, so it is recommended to avoid general anesthesia to allow continuous clinical neurological assessment. The research hypothesis is that rotator cuff repair surgery under LRA alone is possible while maintaining the patient's blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 18 and over
* Patient with a supraspinatus lesion or supraspinatus and infraspinatus lesions requiring surgery for arthroscopic rotator cuff repair, with a non-retracted or minimally retracted tendon (lower stage or = 2 according to the Patte score) and a muscle with little or no fat infiltration (fatty infiltration less than or = 2 according to the Goutallier classification)
* Affiliated participant or beneficiary of a social security scheme.
* Participant having been informed and having given their free, informed and written consent (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patient with a history of surgery for the operated shoulder
* Patient with stage >1 glenohumeral osteoarthritis according to the Samilson classification
* Patient requiring associated subscapularis repair
* Patient with a contraindication to LRA or a contraindication to GA
* Patient wishing a type of anesthesia
* Patient with a contraindication to day surgery
* Patient with neuropathy
* Patients with a history of vagal, emotional or stress-prone discomfort
* Participant whose physical and/or psychological health is severely impaired, which according to the investigator may affect the participant's compliance with the study.
* Patients participating in another research
* Participant in period of exclusion from another research still in progress at the time of inclusion.
* Protected participant: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
* Pregnant, breastfeeding or parturient woman.
* Participant hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
compare systolic blood pressure (SBP) measured during surgery between patients operated for rotator cuff repair under LRA alone and those under LRA and GA. | Day 0
  The main evaluation criterion is the average systolic pressures, measured in the supine position, before loco-regional anesthesia, in the induction room, then in the prone position on entering the operating room, then in a semi-sitting position, and every 5 minutes during the surgery, the duration of which varies according to the patient between 30 and 45 minutes. The average of the systolic blood pressures will be calculated on the available data, with a minimum of 4 values.

SECONDARY OUTCOMES:
Hydraulic pressure during surgery | Day 0
  The difference in pressure administered by the arthrpomp between the beginning and the end of the surgery
The intensity of bleeding during surgery | Day 0
  The intensity of bleeding during surgery, assessed by the number of washes performed
Sedation administered to the patient during surgery | Day 0
  Sedation assessed by the type of sedation administered to the patient: no sedation, hypnotic sedation, morphine sedation
Patient pain after surgery | Day 1 to day 21
  Pain is assessed by a visual analogue scale over 100 mm, measured morning and evening the first 3 days after surgery then once on day 7, day 14 and day 21 after surgery.
Patient satisfaction 3 weeks after surgery | 3 weeks
  Patient satisfaction on the surgery will be measured by a 4 point Likert scale and positive and negative points will be collected in comments
Adverse events between patients operated on LRA alone and patients on LRA and GA. | Day 0 to 6 months
  The number and type of adverse events noted during the procedure and in the 6 months post-operation.
Medication taken for pain between these same groups of patients in the 21 days following surgery. | Day 1 to day 21
  The patient's daily consumption of painkillers will be recorded in a patient diary for 21 days after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BAVEREL, Dr, Principal Investigator — Clinique Bretéché ELSAN
Locations (4):
- France (4):
  - Clinique Bretéché, Nantes
  - CHP St Grégoire, Saint-Grégoire
  - Clinique Belledonne, Saint-Martin-d'Hères
  - Hôpital privé St Claude, Saint-Quentin

IPD SHARING:
Plan to Share IPD: No